CLINICAL TRIAL: NCT05964023
Title: Personalized Brain Functional Sector-guided rTMS Therapy Targeting DLPFC VS "5-centimeter Rule" for Major Depression
Brief Title: pBFS Guided VS "5-cm Rule" rTMS Over DLPFC for MDD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changping Laboratory (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPLMDDDLV5cm
Record Dates: First submitted 2023-07-11; First posted 2023-07-27 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2023-07

CONDITIONS: Major Depression; MDD
Keywords: Major Depression, MDD; pBFS,; 5cm rule
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pBFS rTMS (Experimental): 3 sessions of active rTMS would be delivered to the pBFS-guided left DLPFC daily, with a session of 1800 pulse.
  Interventions: Device: pBFS rTMS
- 5-cm rTMS (Active Comparator): 3 sessions of active rTMS would be delivered to the "5-cm rule" guided left DLPFC daily, with a session of 1800 pulse.
  Interventions: Device: 5-cm rTMS

INTERVENTIONS:
Device: pBFS rTMS — Participants will receive 3 sessions per day of 1800 pulses per session, lasting for 21 days. Individualized targets will be generated using the pBFS method.
  Arms: pBFS rTMS
Device: 5-cm rTMS — Participants will receive 3 sessions per day of 1800 pulses per session, lasting for 21 days. Individualized targets will be localized by "5-cm rule".
  Arms: 5-cm rTMS

SUMMARY:
The investigators aim to investigate whether the intervention effect of pBFS-guided rTMS therapy targeting DLPFC is superior to the intervention effect of the traditional "5 cm-rule" guided rTMS therapy in patients with depressive disorders.

DETAILED DESCRIPTION:
After being informed about the study and potential risks. All patients giving written informed consent will undergo a screening period to determine eligibility for study entry. At week 0, patients who meet the eligibility requirements will be randomized in a blind manner in a 1:1 ratio to the pBFS group, or 5-cm rule group. Then all participants will undergo a 21-day rTMS modulation and 7-day, 14-day, and 45-day post-treatment follow-up visits. Participants will not take any other treatment during the intervention and the 7-day and 14-day post-treatment visits.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria of DSM-5(Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition) for the depression disorder without psychotic symptoms, and currently experiencing recurrence episodes.
* Inpatients or outpatients aged 18-65 years (inclusive), male or female.
* Total HAMD-17 score ≥20 before randomization.Total MADRS score ≥25 before randomization.
* Inadequate response to at least one antidepressant trial of adequate doses and duration.
* Currently not taking any antidepressant medication. If previously medicated, a washout period of 7 days is required.
* Voluntarily participate in the trial and sign informed consent. Able to comply with the planned visit, examination and treatment plan, and other study procedures.

Exclusion Criteria:

* Meet DSM-5 diagnostic criteria for other mental disorders (such as schizophrenia spectrum disorders, bipolar and related disorders, neurodevelopmental disorders, neurocognitive disorders, or depressive disorders due to substances and/or medications, depressive disorders due to other medical problems, etc.);
* Patients with a cardiac pacemaker, cochlear implant, or other metal foreign body and any electronic equipment implanted in the body, patients with claustrophobia and other contraindications to magnetic resonance scanning, and patients with contraindications to rTMS treatment;
* Patients with serious or unstable diseases of the cardiovascular, liver, kidney, blood, endocrine, neurological system, and other systems or organs, especially those with organic brain diseases (such as ischemic stroke, cerebral hemorrhage, brain tumor, etc.) and a history of severe brain trauma as judged by the researcher;
* History of epilepsy (presence of at least 2 uninduced seizures more than 24 hours apart, or diagnosis of the epileptic syndrome, or seizures within the past 12 months); Or currently received medications or other treatments that will lower the seizure threshold;
* History of ECT, rTMS, VNS, DBS, tDCS, light therapy, or other physical therapy related to mental illness within 3 months;
* Currently receiving or planning to start formal cognitive or behavioral therapy, or systemic psychological therapy (interpersonal therapy, dynamic therapy, cognitive behavioral therapy, etc.) during the trial.
* Substance abuse or dependence (including alcohol, drugs, and other psychoactive substances) in the past 1 year;
* The female of childbearing potential plans to become pregnant during the trial and the female that is pregnant or breastfeeding.
* Patients in any clinical trials of other drugs or physical therapy within 1 month before the screening.
* First-degree relatives have bipolar affective disorder.
* There is a significant risk of suicide (MADRS item 10 ≥ 5).
* Difficulty or inability to engage in normal communication, understand or follow instructions, and cooperate with treatment and evaluators.
* Investigators think that was inappropriate to participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-08-20 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Montgomery-Asberg Depression Rating Scale (MADRS) scores | Baseline and Day 21
  The MADRS is a validated instrument stratifying the severity of depressive episodes in adults. The MADRS has an overall score ranging from 0 (no depression) to 60 (worst depression).

SECONDARY OUTCOMES:
changes in MADRS | Baseline, Day 7, Day 14, Day 21 (immediate post-treatment), 7-day post-treatment, 14-day post-treatment, 45-day post-treatment
  The MADRS is a validated instrument stratifying the severity of depressive episodes in adults. The MADRS has an overall score ranging from 0 (no depression) to 60 (worst depression).
changes in HAMD | Baseline, Day 7, Day 14, Day 21 (immediate post-treatment), 7-day post-treatment, 14-day post-treatment, 45-day post-treatment
  The Hamilton Depression Rating Scale (HAMD) is the most widely used clinician-administered depression assessment scale. The HAMD-17 version consists of 17 items，and has an overall score ranging from 0 (no depression) to 52 (worst depression). Higher scores represent higher depression severity.
cognitive change in Digit Symbol Substitution Test (DSST) | Baseline, Day 21 (Immediate Post-treatment)
  Cognitive scores are measured using Chinese brief cognitive test (C-BCT), the DSST equires a subject to match symbols to numbers according to a key located on the top of the page
cognitive change in continuous performance test (CPT) | Baseline, Day 21 (Immediate Post-treatment)
  CPT from the C-BCT measures a person's sustained and selective attention
cognitive change in Trail-Making Test (TMT) | Baseline, Day 21 (Immediate Post-treatment)
  The TMT test from the C-BCT can provide information about visual search speed, scanning, speed of processing, mental flexibility, and executive functioning
cognitive change in Digit Span Test (DST) | Baseline, Day 21 (Immediate Post-treatment)
  DST from the C-BCT is a measure of verbal short term and working memory that can be used in two formats, Forward Digit Span and Reverse Digit Span

CONTACTS AND LOCATIONS:
Overall Officials: Hesheng Liu, Ph.D., Study Chair — Changping Laboratory
Locations (4):
- China (4):
  - Hebei Mental Health Center, Baoding, Hebei
  - Henan Mental Hospital, Xinxiang, Henan
  - Tianjin general hospital, Tianjin, Tianjin Municipality
  - Hangzhou Seventh People's Hospital, Hanzhou, Zhejiang